CLINICAL TRIAL: NCT04182048
Title: Remote Study of an Electronic Means to Characterize Bowel Movements in Adult Populations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HealthMode Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM102001
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome; Healthy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients

SUMMARY:
A remote study to find out if a mobile phone application (HealthMode Stool) can serve as a useful tool to track and characterize daily bowel movements. The application provides participants with a single place to record their bowel movements either as a part of their general health self-monitoring, or because they may be dealing with a bowel movement condition. The minimal study duration is 1 month, and participants can continue using the application up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Females and males over 18 years old
* Willing to use their own/personal mobile phone (iPhone 6 or higher, running iOS 11 or higher) for participation
* Willing to share demographic data with the sponsor of the study
* Willing to follow app use instructions during the course of the study
* Willing to log the bowel movement events on a daily basis with manual input of additional characteristics
* Willing to complete survey instruments as described in study procedures
* Willing to provide electronic informed consent
* Able to read and understand the english language well enough to complete electronic informed consent

Exclusion Criteria:

* New to HealthMode Stool application:
* No additional exclusion criteria.

OR

* Current HealthMode Stool User:
* Is an active participant in any other study using HealthMode Stool app in its protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US resident participants downloading the HealthMode Stool application from the Apple AppStore.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Dataset completeness | 28 days
  Aiming for 90% in two dataset completeness aspects: bowel movement entry days and bowel movement characteristics completeness.

SECONDARY OUTCOMES:
Daily bowel movement characteristics and fluctuation | 28 days
  Measured as category frequency and fluctuations in Bristol Stool Scale items
Daily bowel movement characteristics and fluctuation | 28 days
  Measured as changes in Gastro-intestinal Symptom Rating Scale score. The score ranges from 15 to 105, lower score indicating a better outcome
Daily bowel movement characteristics and fluctuation | 28 days
  Measured as changes in Visceral Sensitivity Index score. The score ranges from 15 to 90, lower score indicating a worse outcome
Usability of the application | 28 days
  Level of usability of the solution by patients by means of a Standard Usability Questionnaire score. The score ranges from 10 to 50, higher score indicating a better usability.

OTHER OUTCOMES:
Sensitivity and specificity of models for automatic determination of bowel movement characteristics | 28 days
  Receiver Operating Characteristic of created mathematical models

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual Facility, The Bronx, New York, United States